CLINICAL TRIAL: NCT06701526
Title: Interventional, Open-label Trial, Investigating the Effectiveness of Eptinezumab in Participants With Migraine and Previous Inadequate Response to CGRP-targeting Therapies
Brief Title: A Trial of Eptinezumab in Participants With Migraine and Insufficient Response to Anti-CGRP Medications
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20668A
Record Dates: First submitted 2024-11-20; First posted 2024-11-22 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Migraine
Keywords: Eptinezumab; CGRP-targeting therapies; anti-CGRP monoclonal antibodies (mAbs); Gepants
MeSH Terms: conditions — Migraine Disorders | interventions — eptinezumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Eptinezumab (Experimental): Participants will receive eptinezumab at Baseline (Day 1) and Week 12
  Interventions: Drug: Eptinezumab

INTERVENTIONS:
Drug: Eptinezumab — Solution for infusion

SUMMARY:
The main goal of this trial is to learn whether eptinezumab improves migraine symptoms and quality of life of participants with migraine who did not perceive a sufficient improvement during previous treatment with therapies targeting calcitonin gene-related peptide (CGRP).

ELIGIBILITY:
Key Inclusion Criteria:

* The participant has a diagnosis of migraine as defined by International Headache Society (IHS) International Classification of Headache Disorders 3rd Edition (ICHD-3) guidelines with a history of migraine of at least 12 months prior to the Screening Visit.
* The participant has ≥8 migraine days per month for each month within the past 3 months prior to the Screening Visit.
* The participant has documented evidence of recent inadequate response to either one anti-CGRP monoclonal antibody (mAb) (other than eptinezumab) or one gepant, indicated and used for migraine prevention.

Key Exclusion Criteria:

* The participant has taken more than 10 tablets of ubrogepant or more than 8 tablets of rimegepant per month as an acute migraine medication in the 1 month prior to the screening visit and during the 4-week baseline period.
* The participant has previously had an inadequate response to more than one CGRP-targeting therapy (anti-CGRP mAb or gepants), indicated for migraine prevention.
* The participant has a history of cancer, other than basal cell or stage 1 squamous cell carcinoma of the skin or adequately treated cervical intraepithelial neoplasia, that has not been in remission for >5 years prior to the first dose of eptinezumab. Male participants with abnormal prostate-specific antigen levels according to national/local guideline may be enrolled in the trial provided they have been followed up, have been asymptomatic, and have had no treatment for prostate cancer. Participants under surveillance for a low and stable level of M-component are allowed.
* The participant has previously been treated with eptinezumab.

Other protocol-defined inclusion and exclusion criteria apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-12-18 (Actual); Primary Completion 2026-06-05 (Estimated); Study Completion 2026-06-05 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Response of "Much Improved" or "Very Much Improved" on the Patient Global Impression of Change (PGIC) Scale | Week 24

SECONDARY OUTCOMES:
Change from Baseline in Monthly Migraine Days (MMDs) | Weeks 1-12 and 13-24
Change from Baseline in the Percentage of MMDs with Severe Pain Intensity | Weeks 1-12 and 13-24
Change from Baseline in Monthly Headache Days (MHDs) | Weeks 1-12 and 13-24
Change from Baseline in MMDs with Use of Acute Medication | Weeks 1-12 and 13-24
Number of Participants with Response of "Much Improved" or "Very Much Improved" on the PGIC Scale | Week 12
PGIC Score | Weeks 12 and 24
Change from Baseline in Migraine Disability Assessment (MIDAS) Scores | Weeks 12 and 24
Goal Attainment Scaling (GAS) Score | Weeks 12 and 24
Number of Participants with GAS Score ≥50 | Weeks 12 and 24
Change from Baseline in Number of Good Days per Month | Weeks 12 and 24
Change from Baseline in Migraine Clinical Outcome Assessment System-Cognition (MiCOAS-COG) Score | Weeks 12 and 24
Number of Participants with Response of "Much Improved" or "Very Much Improved" in Brain Fog | Weeks 12 and 24
Brain Fog Score | Weeks 12 and 24
Number of Participants with Response of "Much Improved" or "Very Much Improved" on the Clinical Global Impression of Change (CGIC) Scale | Weeks 12 and 24
CGIC Score | Weeks 12 and 24
Number of Participants with Adverse Events (AEs) | Up to Week 26

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — HQ_Medinfo@Lundbeck.com
Locations (28):
- United States (28):
  - Neuropain Medical Center, Fresno, California
  - Sunwise Clinical Research, LLC., Oakland, California
  - The Neuron Clinic, San Marcos, California
  - St. Joseph's Hospital and Medical Center - Barrow Neurological Institute, Aurora, Colorado
  - Advanced Neurology of Colorado, LLC, Longmont, Colorado
  - Research of the Rockies, Parker, Colorado
  - Hasbani & Hasbani MDs, New Haven, Connecticut
  - New England Institute for Neurology and Headache, Stamford, Connecticut
  - Brainstorm Research, Miami, Florida
  - Premiere Research Institute at Palm Beach Neurology, West Palm Beach, Florida
  - PANDA Neurology and Atlanta Headache Specialists, Atlanta, Georgia
  - St Luke's Meridian Medical Center, Meridian, Idaho
  - Chicago Headache Center & Research Institute, Chicago, Illinois
  - Crescent City Headache and Neurology, New Orleans, Louisiana
  - Neurology Center of New England P.C., Foxborough, Massachusetts
  - MedVadis Research Corporation, Watertown, Massachusetts
  - Mass Institute of Clinical Research, Westborough, Massachusetts
  - Memorial Healthcare, Owosso, Michigan
  - Albany Medical College, Albany, New York
  - Dent Neurosciences Research Center, Inc., Amherst, New York
  - North Suffolk Neurology, Port Jefferson Station, New York
  - NeuroScience Research Center, LLC., Canton, Ohio
  - C7 Research, Cleveland, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Preferred Primary Care Physicians, Inc., Pittsburgh, Pennsylvania
  - KCA Neurology, PLLC, Franklin, Tennessee
  - Texas Neurology, PA, Dallas, Texas
  - Inova Health Care Services, Fairfax, Virginia